CLINICAL TRIAL: NCT04952662
Title: Candidate Gene Association Study With Injury, Non-Contact Injury, Non-Contact Muscle Injury, Fracture and Apophysitis Injury in Elite Male Youth Football Players
Brief Title: Candidate Gene Association Study With Injury in Elite Male Youth Football Players
Status: Completed | Type: Observational
Sponsor: St Mary's University College (Other)
Collaborators: Fulham Football Club (Unknown)
Responsible Party: Sponsor
Other Study IDs: SMEC_2019-20_002
Record Dates: First submitted 2021-05-31; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Injuries; Genetic Change
Keywords: SNP; Apophysitis; Fracture; Strain; Sprain; Genetic; Injury
MeSH Terms: conditions — Wounds and Injuries; Fractures, Bone; Sprains and Strains | interventions — Pharmacogenomic Variants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Genetic variants — COL1A1 rs1800012, COL1A2 rs412777, COL5A1 rs12722, ACTN3 rs1815739, ACE rs1799752, ESR1 rs2234693, MMP3 rs679620, VDR rs2228570 and GDF5 rs143383

SUMMARY:
Understanding how candidate genes, previously associated with injury susceptibility, influence the incidence of muscle, bone, ligament, and tendon injuries across the development pathway of elite footballers may provide valuable insight into inherent injury predisposition to support the long-term development of every individual. Therefore, the aim of the present study was to investigate the association between candidate genetic variants and muscle, bone, ligament, and tendon injuries in elite football with sub-analysis of the influence of age and maturation on injury susceptibility.

DETAILED DESCRIPTION:
Genetic variants in several candidate genes which code for structural constituents (COL1A1 rs1800012, COL1A2 rs412777, COL5A1 rs12722 and ACTN3 rs1815739), regulatory components (ACE rs1799752, ESR1 rs2234693 and MMP3 rs679620) and transcription factors (VDR rs2228570 and GDF5 rs143383) affecting the form, function and injury susceptibility of muscle, bone, ligament, and tendon tissue will be associated with overall injury, non-contact, bone, ligament, tendon and apophysitis injury risk in elite male youth and adult footballers.

ELIGIBILITY:
Inclusion Criteria:

* Elite Male Footballer Player Registered at Fulham Football Club

Exclusion Criteria:

* Female no longer registered at Fulham Football Club

Ages: 8 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Elite male youth football players
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of non-injured and injured participants with injury risk alleles | 8 Years
  Injury, Non-Contact Injury, Non-Contact Muscle Injury, Fracture and Apophysitis Injury

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Fulham Football Club, London, New Malden
  - St Mary's University, Twickenham, London, Twickenham

IPD SHARING:
Plan to Share IPD: No